CLINICAL TRIAL: NCT04161651
Title: Evaluation of Long-Term Implanted Sensor in Patients on Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: DYN Diagnostic LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0047-19-COM
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes
Keywords: eversense; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental)
  Interventions: Device: eversense

INTERVENTIONS:
Device: eversense — eversense CGM

SUMMARY:
Evaluation of Long-Term Implanted Sensor in Patients on Quality of life

DETAILED DESCRIPTION:
Assess satisfaction and acceptance of long-term implanted single sensor use (eversense XL) for up to 6 months in type 1 insulin-using patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female diagnosed with type 1 diabetes mellitus
2. Age > 18
3. Insulin treatment for at least 1 year (Either MDI of CSII)
4. HbA1c < 11%
5. Signing informed consent and willing to apply with study procedure

Exclusion Criteria:

1. History of severe hypoglycaemia in the last 3 months
2. History of DKA in the last 3 months
3. Any condition preventing or complicating the placement, operation or removal of the Sensor including upper extremity deformities or skin condition
4. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study
5. Any condition that require MRI imaging or planned MRI during the trial period
6. Known topical or local anaesthetic allergy
7. Known allergy to glucocorticoids
8. History of hepatitis B, hepatitis C or HIV
9. Any Bleeding disorder or taking anticoagulant medication
10. Participation in other clinical trial
11. Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
changes in quality of life evaluated questionnaires (DTSQ) | 6 months

SECONDARY OUTCOMES:
Change in HBA1C | 3 / 6 months
CGM Time In Range (70-180 mg/dl) | 3 / 6 months
CGM Time in hypoglycaemia below 70 mg/dl | 3 / 6 months
CGM Time in hypoglycaemia below 54 mg/dl | 3 / 6 months
CGM time in range difference [2 weeks before digital visit and 2 weeks after digital visit] | 3 / 6 months
Change in HFS-ii (hypoglycaemia fear survey II) | 6 months
Change in Continuous Glucose Monitor Satisfaction Scale (CGM-SAT) | 6 months
Any adverse event related to study device | 6 months

IPD SHARING:
Plan to Share IPD: No